CLINICAL TRIAL: NCT00712439
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Gabapentin Extended Release (G-ER) Tablets in the Treatment of Patients With Painful Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy of Gabapentin in Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Lynne Rowe, Depomed
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81-0046
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: DPN,; Diabetic; Peripheral; Neuropathy; Painful
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Gabapentin Extended Release tablets
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin Extended Release tablets
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a new Gabapentin tablet, is safe and effective for the treatment of painful diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years or older with diagnosis of type 1 or type 2 diabetes who have reported symmetrical painful symptoms in distal extremities for 1-5 years prior to the study and whose symptoms are attributable to sensorimotor diabetic peripheral neuropathy (DPN).
* Patients of childbearing potential must have a negative urine pregnancy test at screening/randomization, and must use medically acceptable methods of birth control.
* Patient has pain score of at least 4 on the 11-point Likert numerical rating scale at screening. Potential patients should not be informed of the pain intensity eligibility criterion prior to screening or randomization.
* Patient has a mean baseline week pain intensity of at least 4 on the 11-point Likert scale at the end of a one-week pre-treatment period and has completed at least 4 days of diary entries during the baseline week.
* Patient is on stable regimen of antidiabetes medication at screening that can be maintained during the study.
* Patient has hemoglobin A1c (HbA1c) ≤11% at screening.
* Patient has FPG ≤310 mg/dL at screening.
* Patient must have a minimum washout of greater than 5 times the half-life of the drug of any of several medications
* Patients currently treated with gabapentin or pregabalin at screening may be eligible for the study, but must have tapering period wherein the dose of gabapentin is reduced gradually over a period of at least 7 days plus a 2-day or 3-day washout of gabapentin or pregabalin, respectively, prior to start of the Baseline Week.
* Patient must have adequate eyesight to complete questions on the DiaryPro and SitePro. If a patient is unable to do so (for reasons other than severe eye disease) but a caregiver is available to complete these tasks following instruction from the patient, the caregiver may be trained to accomplish these tasks

Exclusion Criteria:

* Patients who have previously not responded to treatment for DPN with gabapentin at doses of ≥1200 mg/day or pregabalin at doses ≥300 mg/day.
* Patients who previously experienced dose-limiting adverse effects that prevented titration of gabapentin to an effective dose.
* Patient has hypersensitivity to gabapentin.
* Patient is a nursing mother.
* Patient has used injected anesthetics or steroids within 30 days of baseline.
* Patient has certain conditions that could confound evaluation of painful DPN, in particular, amputations other than toes, non-diabetic neurologic disorders (e.g. phantom limb pain), and skin conditions affecting sensation in painful limbs.
* Patient has skin conditions in the area affected by the neuropathy that could alter sensation.
* Patient is in an immunocompromised state.
* Patient has an estimated creatinine clearance of <60 ml/min calculated using the Cockroft Gault method (Appendix 3).
* Patient has had malignancy within past 2 years other than basal cell carcinoma.
* Patient has had gastric reduction surgery.
* Patient has severe chronic diarrhea, chronic constipation [unless attributed to drugs that will be washed out], uncontrolled irritable bowel syndrome (IBS) or unexplained weight loss.
* Patient has any abnormal chemistry or hematology results that are deemed by the investigator to be clinically significant.
* Patient has a history of substance abuse within the past year.
* Patient has had 1 or more visits to an emergency room or hospital within the previous 30 days due to hypoglycemia.
* Patient has a history of seizure (except for infantile febrile seizure) or is at risk of seizure due to head trauma.
* Patient has a history of pernicious anemia, untreated hypothyroidism, chronic hepatitis B or C, hepatitis within the past 3 months, or HIV infection.
* Patient has any other serious medical condition that, in the opinion of the Investigator would jeopardize the safety of the patient or affect the validity of the study results.
* Continuing use of any concomitant medication excluded by Inclusion Criterion 8.
* Patient has participated in a clinical trial of an investigational drug or device within 30 days of the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary study objective is to assess the relative efficacy of G-ER versus placebo in reducing the mean daily pain score from the baseline week to end of efficacy treatment period (Treatment Week 4) in patients with DPN. | 4 weeks

SECONDARY OUTCOMES:
Secondary efficacy measures will include changes from baseline in average daily sleep interference scores, SF-MPQ, BPI,NPS, PGIC, and CGIC. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sathyanarayana, Study Director — Depomed

REFERENCES:
- [Derived] Sandercock D, Cramer M, Biton V, Cowles VE. A gastroretentive gabapentin formulation for the treatment of painful diabetic peripheral neuropathy: efficacy and tolerability in a double-blind, randomized, controlled clinical trial. Diabetes Res Clin Pract. 2012 Sep;97(3):438-45. doi: 10.1016/j.diabres.2012.03.010. Epub 2012 Apr 11. PMID 22497967
- [Derived] Sandercock D, Cramer M, Wu J, Chiang YK, Biton V, Heritier M. Gabapentin extended release for the treatment of painful diabetic peripheral neuropathy: efficacy and tolerability in a double-blind, randomized, controlled clinical trial. Diabetes Care. 2009 Feb;32(2):e20. doi: 10.2337/dc08-1450. No abstract available. PMID 19171730